CLINICAL TRIAL: NCT01684930
Title: Increased Plasma Nitrite, Tissue Oxygenation and Functional Changes in PAD
Brief Title: Nitrites, Exercise, and Peripheral Arterial Disease
Acronym: NO-PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason Allen, Ph.D., Assistant Professor Doctor of Physical Therapy Program & Division of Cardiovascular Medicine, Duke University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00031918; 1R21HL111972-01 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Cardiovascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Exercise; Functional Capacity
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BR Juice (Beet-It Stamina Shot) and Exercise Training (Experimental): Subjects consume 70 ml of Beetroot Juice (Beet-It Stamina Shot) to assess acute effects of beverage supplementation at the start (between Testing Visits 1 & 2) and at the end of the trial (between Visits 3 & 4). It also allows for comparisons of the combination of beetroot juice and chronic training effects (between Visits 2 & 3) to when the subject has not consumed the beverage (Visits 1 & 4). All subjects will consume Beet-It Stamina Shot 3 hours prior to all beverage tolerance visits, Testing Visits 2 & 3 and for all supervised exercise training visits during the 12 week intervention.
  Interventions: Drug: Beetroot Juice (Beet-It Stamina Shot) & Supervised Exercise Training
- BR Juice Placebo and Exercise Training (Placebo Comparator): Subjects consume 70 ml of Beetroot Juice (Beet-It Stamina Shot; Placebo) to assess acute effects of beverage supplementation at the start (between Testing Visits 1 & 2) and at the end of the trial (between Visits 3 & 4). It also allows for comparisons of the combination of placebo beverage and chronic training effects (between Visits 2 & 3) to when the subject has not consumed the beverage (Visits 1 & 4). All subjects will consume Beet-It Stamina Shot (Placebo) 3 hours prior to all beverage tolerance visits, Testing Visits 2 & 3 and for all supervised exercise training visits during the 12 week intervention.
  Interventions: Other: Placebo Comparator Beverage (Beet-It Stamina Shot) & Exercise Training

INTERVENTIONS:
Drug: Beetroot Juice (Beet-It Stamina Shot) & Supervised Exercise Training — The beverage is high in inorganic nitrate and bottled and supplied by James White Drinks. This supplement will be used in conjunction with supervised exercise training.
  Other Names: James White Drinks
  Arms: BR Juice (Beet-It Stamina Shot) and Exercise Training
Other: Placebo Comparator Beverage (Beet-It Stamina Shot) & Exercise Training — The beverage is identical in look and taste to Beet-It Stamina Shot but with active ingredient removed. It is also bottled and supplied by James White Drinks. This placebo supplement will be used in conjunction with supervised exercise training.
  Other Names: James White Drinks
  Arms: BR Juice Placebo and Exercise Training

SUMMARY:
The hypothesis of this proposal is that in subjects with PAD, regular consumption of a high nitrate supplement which raises plasma nitrite, in conjunction with 12 weeks of supervised exercise training at the limb ischemic threshold (SET) will produce a greater clinical benefit (increases in COT and PWT) than placebo plus supervised exercise at the limb ischemic threshold (PET).

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Arterial Disease (ABI of less than 0.9)
* Intermittent Claudication for 3 or more months

Exclusion Criteria:

* Individuals with known alcohol or drug abuse problems
* Individuals who have suffered a heart attack or stroke, or have changes on a resting ECG, in the last 3 months
* Those classified as American Heart Association Class D
* Gangrene, impending limb loss or osteomyelitis
* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment
* Severe peripheral neuropathy
* Any condition other than PAD that limits walking
* Chest pain during treadmill exercise which appears before the onset of claudication, or >3mm ST depression during exercise
* Subjects taking nitrates or nitroglycerin products
* Must not be taking protein pump inhibitor medications

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Diet & Fitness Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Woessner M, VanBruggen MD, Pieper CF, Sloane R, Kraus WE, Gow AJ, Allen JD. Beet the Best? Circ Res. 2018 Aug 31;123(6):654-659. doi: 10.1161/CIRCRESAHA.118.313131. PMID 29976553
- [Derived] Woessner MN, VanBruggen MD, Pieper CF, O'Reilly EK, Kraus WE, Allen JD. Combined Dietary Nitrate and Exercise Intervention in Peripheral Artery Disease: Protocol Rationale and Design. JMIR Res Protoc. 2017 Oct 3;6(10):e139. doi: 10.2196/resprot.7596. PMID 28974486
- See also: Frederick R. Cobb Non-Invasive Vascular Research Laboratory — http://cardiology.medicine.duke.edu/research/clinical-research/frederick-r-cobb-non-invasive-vascular-research-laboratory
- See also: Duke Clinical Trials Listing — http://www.dukehealth.org/clinicaltrials/20120705125024398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10,817 patients were screened, 898 potential study candidates were identified, and 32 subjects signed consent and were enrolled from June 2012 through July 2014. Of the 32 subjects who signed consent, 5 subjects were screen failures and 1 withdrew consent. 26 subjects were randomized and 22 subjects completed all study testing.
Period: Overall Study
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Started | 12 | 14
Completed | 9 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.25 (8.9) | 71.85 (7.9) | 67.88 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity: VO2peak (Maximal Oxygen Consumption)
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test with expired gas analysis, for determination of peak oxygen consumption, claudication onset time and peak walking time.
Time Frame: Baseline and 16 Weeks
Population: All participants who completed study.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 9 | 13
ml/kg/min | 1.48 (2.69) | 0.23 (2.21)

2. Primary Outcome: Change In Time To Exhaustion
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test with expired gas analysis, for determination of total time to exhaustion.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 9 | 13
seconds | 289.56 (175.44) | 254.92 (210.48)

3. Secondary Outcome: Change in Functional Ability
Description: Six-Minute Walk test. This test simple and practical assessment of functional capacity. The test measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes. The test is self-paced and assesses the submaximal level of functional capacity. The subjects choose their own intensity and are allowed to stop and rest if necessary during the test.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 9 | 13
feet | 172.89 (166.05) | 95 (173.7)

4. Secondary Outcome: Change In Claudication Onset Time
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test with expired gas analysis, for determination of claudication onset time.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 9 | 13
seconds | 199.22 (143.47) | 48.58 (198.75)

5. Secondary Outcome: Change In Vascular Function (BAFMD)
Description: Vascular Function is measured as Brachial artery flow-mediated dilation (BAFMD). BAFMD is a measure of change in artery diameter after a stimulus .
Time Frame: Baseline and 16 weeks
Population: participants with analyzable data
Measure: Mean (Standard Deviation); unit: % dilation
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 4 | 6
% dilation | -1.14 (3.02) | -0.19 (1.80)

6. Secondary Outcome: Change in Angiogenesis
Description: Gastrocnemious muscle biopsy will be performed to measure the number of capillaries per fibre as a marker of change in angiogenesis between groups
Time Frame: Baseline and 16 weeks
Population: Participants who had a gastrocnemius muscle biopsy with enough tissue to analyze.
Measure: Mean (Standard Deviation); unit: capillaries per fibrer
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 8
capillaries per fibrer | 0.38 (0.54) | 0.26 (0.51)

ADVERSE EVENTS:
Arm/Group | BR Juice (Beet-It Stamina Shot) and Exercise Training | BR Juice Placebo and Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 1/12 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BR Juice (Beet-It Stamina Shot) and Exercise Training (N=12) | BR Juice Placebo and Exercise Training (N=14)
hypotensive episode with exercise (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The largest limitation to the study was the evolving knowledge on conversion rates of oral inorganic nitrate to nitrite. We found a good deal of unexpected inter and intra-subject variation in conversion rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes